CLINICAL TRIAL: NCT04157686
Title: A Multicenter, Long-term, Open-label Study to Evaluate the Safety of MT10109L (NivobotulinumtoxinA) for the Treatment of Glabellar Lines and Lateral Canthal Lines
Brief Title: MT10109L in the Long-term, Open-label Treatment of Glabellar Lines (GL) and Lateral Canthal Lines (LCL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT10109L-004; 2014-005303-24 (EudraCT Number)
Record Dates: First submitted 2019-10-23; First posted 2019-11-08 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Glabellar Lines; Lateral Canthal Lines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (8):
- Placebo/MT10109L Dose 1 (Experimental): The participant pool in this arm are from the MT10109L-001 lead-in study (NCT03795922), who received Placebo in period 1 and MT10109L Dose 1 in period 2. Eligible participants from this study continue receiving Dose 1 in the open-label MT10109L-004 study
  Interventions: Drug: MT10109L Dose 1
- Placebo/MT10109L Dose 2 (Experimental): The participant pool in this arm are from the MT10109L-002 lead-in study (NCT03785145), who received Placebo in period 1 and MT10109L Dose 2 in period 2. Eligible participants from this study continue receiving Dose 2 in the open-label MT10109L-004 study.
  Interventions: Drug: MT10109L Dose 2
- Placebo/MT10109L Dose 1 + Dose 2 (Experimental): The participant pool in this arm are from the MT10109L-005 (NCT03721016) and MT10109L-006 (NCT03732833) lead-in studies, who received Placebo in periods 1 & 2. Eligible participants from this study receives Dose 1 into the GL area and Dose 2 into the LCL area in the open-label MT10109L-004 study.
  Interventions: Drug: MT10109L Dose 1 + Dose 2
- MT10109L Dose 1/Dose 1 (Experimental): The participant pool in this arm are from the MT10109L-001 lead-in study (NCT03795922), who received MT10109L Dose 1 each in period 1 and period 2. Eligible participants from this study continue receiving Dose 1 in the open-label MT10109L-004 study.
  Interventions: Drug: MT10109L Dose 1
- MT10109L Dose 2/Dose 2 (Experimental): The participant pool in this arm are from the MT10109L-002 lead-in study (NCT03785145), who received MT10109L Dose 2 each in period 1 and period 2. Eligible participants from this study continue receiving Dose 2 in the open-label MT10109L-004 study.
  Interventions: Drug: MT10109L Dose 2
- MT10109L Dose 1/Dose 1+2 (Experimental): The participant pool in this arm are from the from MT10109L-005 lead-in study (NCT03721016), who received MT10109L Dose 1 in periods 1 and 2. Eligible participants from this study receives Dose 1 into the GL area and Dose 2 into the LCL area in the open-label MT10109L-004 study.
  Interventions: Drug: MT10109L Dose 1 + Dose 2
- MT10109L Dose 2/Dose 1+2 (Experimental): The participant pool in this arm are from the MT10109L-006 lead-in study (NCT03732833), who received MT10109L Dose 2 in periods 1 and 2. Eligible participants from this study receives Dose 1 into the GL area and Dose 2 into the LCL area in the open-label MT10109L-004 study.
  Interventions: Drug: MT10109L Dose 1 + Dose 2
- MT10109L Dose 1+2/Dose 1+2 (Experimental): The participant pool in this arm are from the MT10109L-005 (NCT03721016) and MT10109L-006 (NCT03732833) lead-in studies, who received MT10109L Dose 1 into GL and Dose 2 into LCL in periods 1 & 2. Eligible participants from this study receives Dose 1 into the GL area and Dose 2 into the LCL area in the open-label MT10109L-004 study.
  Interventions: Drug: MT10109L Dose 1 + Dose 2

INTERVENTIONS:
Drug: MT10109L Dose 1 — MT10109L Dose 1 will be injected into the GL area
  Arms: MT10109L Dose 1/Dose 1; Placebo/MT10109L Dose 1
Drug: MT10109L Dose 2 — MT10109L Dose 2 will be injected into the LCL area
  Arms: MT10109L Dose 2/Dose 2; Placebo/MT10109L Dose 2
Drug: MT10109L Dose 1 + Dose 2 — MT10109L Dose 1 will be injected into the GL area plus MT10109L Dose 2 will be injected into the LCL area
  Arms: MT10109L Dose 1+2/Dose 1+2; MT10109L Dose 1/Dose 1+2; MT10109L Dose 2/Dose 1+2; Placebo/MT10109L Dose 1 + Dose 2

SUMMARY:
To evaluate the long-term safety of MT10109L in the treatment of GL and/or LCL in participants with moderate to severe GL and/or LCL.

DETAILED DESCRIPTION:
Study MT10109L-004 is an open-label extension involving participants from studies MT10109L-001 (NCT03795922), -002 (NCT03785145), -005 (NCT03721016), and -006 (NCT03732833) (referred to as Lead-In studies). The objective is to evaluate long term safety of MT10109L. Participants will include those who completed the global lead-in studies and meet the eligibility criteria for entering this open-label extension study.

Participants who meet retreatment criteria will receive MT10109L administered in the same treatment area(s) with the same number of injections and injection sites as in their lead-in studies.

The safety and efficacy data from the lead-in and this open-label extension will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* Completion of lead-in Phase 3 study;
* Female participants must not be pregnant or planning to get pregnant and willing to minimize the risk of inducing pregnancy for the duration of the clinical study and follow-up period.

Exclusion Criteria:

* Known immunization or hypersensitivity to any botulinum toxin serotype;
* Any medical condition that may put the participant at increased risk with exposure to MT10109L including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other condition that might interfere with neuromuscular function;
* Known allergy or sensitivity to any of the components of the study interventions, or any materials used in the study procedures;
* Females who are pregnant, nursing, or planning a pregnancy during the study;
* Participants who plan for an extended absence away from the immediate area of the study site that would preclude them from returning for all protocol-specified study visits.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 957 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SangMi Park, Study Director — Medytox Inc.
Locations (38):
- United States (18):
  - Clear Dermatology & Aesthetics Center, Scottsdale, Arizona
  - The Eye Research Foundation, Newport Beach, California
  - Art of Skin MD, Solana Beach, California
  - Susan H. Weinkle, Bradenton, Florida
  - Skin Research Institute, Coral Gables, Florida
  - Coleman Center For Cosmetic Dermatologic Surgery, Metairie, Louisiana
  - Etre Cosmetic Dermatology and Laser Center, New Orleans, Louisiana
  - MD Laser Skin & Vein, Hunt Valley, Maryland
  - Laser & Skin Surgery Center of New York, New York, New York
  - Skin Search of Rochester Inc., Rochester, New York
  - M3 Wake Research Inc., Raleigh, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Aventiv Research Dublin, Dublin, Ohio
  - Westlake Dermatology & Cosmetic Surgery - Westlake, Austin, Texas
  - DermResearch Inc., Austin, Texas
  - Bellaire Dermatology, Bellaire, Texas
  - SkinDC, Arlington, Virginia
  - Virginia Clinical Research, Inc., Norfolk, Virginia
- Belgium (2):
  - UZ Brussel, Jette, Brussels Capital
  - Medical Skincare, Sint-Truiden, Limburg
- Canada (6):
  - Dr. Shannon Humphrey Inc., Vancouver, British Columbia
  - Project Skin MD LTD, Vancouver, British Columbia
  - Pacific Derm, Vancouver, British Columbia
  - Dermetics Cosmetic Dermatology, Burlington, Ontario
  - The Center For Dermatology, Richmond Hill, Ontario
  - Sweat Clinics of Canada, Toronto, Ontarion
- Germany (5):
  - Rosenpark Research, Darmstadt
  - Privatpraxis Dr. Hilton & Partner, Düsseldorf
  - Hautok and Hautok-cosmetics, München
  - Studienzentrum Theatiner46, München
  - MediCorium Zentrum fuer Dermatologie und Aesthetik, Oberursel
- Russia (4):
  - Kazan State Medical University, Kazan'
  - Medical Center Capital - Zdorovie LLC, Moscow
  - Center dermatovenereology and cosmetology, Moscow
  - State Budget Institution of Higher Education North, Saint Petersburg
- United Kingdom (3):
  - Meyer Clinic, Chichester
  - NHS Lanarkshire, Glasgow
  - MediZen Premier Aesthetic Clinic, Sutton Coldfield

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approximately 800 participants were planned to be enrolled. A total of 957 participants were enrolled and treated, and 759 participants completed the study. There were 957 participants in the intent-to-treat (ITT) population, which were used for the efficacy of US FDA and safety analyses.
Pre-assignment Details: Study MT10109L-004 is an open-label extension involving participants from studies MT10109L-001 (NCT03795922), -002 (NCT03785145), -005 (NCT03721016), and -006(NCT03732833) (referred to as Lead-In studies). Participants from the lead-in studies, who met the eligibility criteria, were enrolled to continue receiving additional cycles of MT10109L in their respective treatment areas (Glabellar area or Lateral Canthal Lines area).
Groups:
- Placebo/MT10109L Dose 1: The participant pool in this arm were from the MT10109L-001 lead-in study (NCT03795922), who received Placebo in period 1 and MT10109L Dose 1 in period 2. Eligible participants from this study continued receiving Dose 1 in the open-label MT10109L-004 study
  MT10109L Dose 1: MT10109L Dose 1 was injected into the GL area.
- Placebo/MT10109L Dose 2: The participant pool in this arm were from the MT10109L-002 lead-in study (NCT03785145), who received Placebo in period 1 and MT10109L Dose 2 in period 2. Eligible participants from this study continued receiving Dose 2 in the open-label MT10109L-004 study.
  MT10109L Dose 2: MT10109L Dose 2 was injected into the LCL area.
- Placebo/MT10109L Dose 1 + Dose 2: The participant pool in this arm were from the MT10109L-005 (NCT03721016) and MT10109L-006 (NCT03732833) lead-in studies, who received Placebo in periods 1 & 2. Eligible participants from this study received Dose 1 into the GL area and Dose 2 into the LCL area in the open-label MT10109L-004 study.
  MT10109L Dose 1 + Dose 2: MT10109L Dose 1 was injected into the GL area plus MT10109L Dose 2 was injected into the LCL area.
- MT10109L Dose 1/Dose 1: The participant pool in this arm were from the MT10109L-001 lead-in study (NCT03795922), who received MT10109L Dose 1 each in period 1 and period 2. Eligible participants from this study continued receiving Dose 1 in the open-label MT10109L-004 study.
  MT10109L Dose 1: MT10109L Dose 1 was injected into the GL area
- MT10109L Dose 2/Dose 2: The participant pool in this arm were from the MT10109L-002 lead-in study (NCT03785145), who received MT10109L Dose 2 each in period 1 and period 2. Eligible participants from this study continued receiving Dose 2 in the open-label MT10109L-004 study.
  MT10109L Dose 2: MT10109L Dose 2 was injected into the LCL area.
- MT10109L Dose 1/Dose 1+2: The participant pool in this arm were from the from MT10109L-005 lead-in study (NCT03721016), who received MT10109L Dose 1 in periods 1 and 2. Eligible participants from this study received Dose 1 into the GL area and Dose 2 into the LCL area in the open-label MT10109L-004 study.
  MT10109L Dose 1 + Dose 2: MT10109L Dose 1 was injected into the GL area plus MT10109L Dose 2 was injected into the LCL area.
- MT10109L Dose 2/Dose 1+2: The participant pool in this arm were from the MT10109L-006 lead-in study (NCT03732833), who received MT10109L Dose 2 in periods 1 and 2. Eligible participants from this study received Dose 1 into the GL area and Dose 2 into the LCL area in the open-label MT10109L-004 study.
  MT10109L Dose 1 + Dose 2: MT10109L Dose 1 was injected into the GL area plus MT10109L Dose 2 was injected into the LCL area
- MT10109L Dose 1+2/Dose 1+2: The participant pool in this arm were from the MT10109L-005 (NCT03721016) and MT10109L-006 (NCT03732833) lead-in studies, who received MT10109L Dose 1 into GL and Dose 2 into LCL in periods 1 & 2. Eligible participants from this study received Dose 1 into the GL area and Dose 2 into the LCL area in the open-label MT10109L-004 study.
  MT10109L Dose 1 + Dose 2: MT10109L Dose 1 was injected into the GL area plus MT10109L Dose 2 was injected into the LCL area.
Period: Overall Study
Arm/Group | Placebo/MT10109L Dose 1 | Placebo/MT10109L Dose 2 | Placebo/MT10109L Dose 1 + Dose 2 | MT10109L Dose 1/Dose 1 | MT10109L Dose 2/Dose 2 | MT10109L Dose 1/Dose 1+2 | MT10109L Dose 2/Dose 1+2 | MT10109L Dose 1+2/Dose 1+2
Started | 55 | 56 | 118 | 116 | 108 | 128 | 123 | 253
Completed | 43 | 41 | 89 | 87 | 83 | 106 | 92 | 218
Not Completed | 12 | 15 | 29 | 29 | 25 | 22 | 31 | 35
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 3 | 0 | 0 | 0 | 3 | 0
Not completed — Lost to Follow-up | 1 | 2 | 8 | 6 | 6 | 3 | 7 | 9
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 10 | 10 | 12 | 20 | 12 | 11 | 18 | 24
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — COVID-19, Family Reasons etc. | 0 | 2 | 4 | 1 | 4 | 6 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants pool in this open-label extension study flowed from studies MT10109L-001 (NCT03795922), -002 (NCT03785145), -005 (NCT03721016), and -006 (NCT03732833) (referred to as Lead-In studies). 957 participants were included in the Intent-To-Treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/MT10109L Dose 1 | Placebo/MT10109L Dose 2 | Placebo/MT10109L Dose 1 + Dose 2 | MT10109L Dose 1/Dose 1 | MT10109L Dose 2/Dose 2 | MT10109L Dose 1/Dose 1+2 | MT10109L Dose 2/Dose 1+2 | MT10109L Dose 1+2/Dose 1+2 | Total
Number analyzed (Participants) | 55 | 56 | 118 | 116 | 108 | 128 | 123 | 253 | 957
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 54 | 110 | 107 | 103 | 120 | 113 | 241 | 902
  >=65 years | 1 | 2 | 8 | 9 | 5 | 8 | 10 | 12 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (10.18) | 46.7 (11.75) | 48.2 (11.68) | 46.9 (12.17) | 47.1 (10.34) | 47.8 (11.24) | 48.5 (10.53) | 47.9 (10.80) | 47.7 (11.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 42 | 99 | 106 | 87 | 109 | 103 | 227 | 826
  Male | 2 | 14 | 19 | 10 | 21 | 19 | 20 | 26 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 12 | 3 | 17 | 19 | 5 | 23 | 85
  Not Hispanic or Latino | 54 | 51 | 106 | 113 | 91 | 109 | 118 | 230 | 872
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 5
  Asian | 1 | 1 | 1 | 1 | 4 | 3 | 3 | 4 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 1 | 2 | 3 | 3 | 2 | 1 | 1 | 4 | 17
  White | 53 | 53 | 113 | 112 | 101 | 123 | 119 | 241 | 915
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Any Adverse Event (AE)
Description: The safety analyses were conducted in the Intent-to-Treat (ITT) population. All adverse events were collected from the signing of the ICF to 30 days after the participant's last study visit.
Time Frame: Baseline to Day 720 or Study Exit
Population: All safety analyses were carried out using the ITT population, which was defined as all participants who enrolled in Study MT10109L-004 and received at least 1 intervention (MT10109L or placebo) in their prior Phase 3 study (MT10109L-001, -002, -005, or -006) or in the current study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/MT10109L Dose 1 | Placebo/MT10109L Dose 2 | Placebo/MT10109L Dose 1 + Dose 2 | MT10109L Dose 1/Dose 1 | MT10109L Dose 2/Dose 2 | MT10109L Dose 1/Dose 1+2 | MT10109L Dose 2/Dose 1+2 | MT10109L Dose 1+2/Dose 1+2
Number analyzed (Participants) | 55 | 56 | 118 | 116 | 108 | 128 | 123 | 253
Participants | 39 | 39 | 80 | 89 | 74 | 80 | 89 | 183

2. Primary Outcome: Number of Participants Who Experienced Treatment-Related Adverse Events (TEAEs)
Description: This section focuses primarily on Treatment-Related (Study drug or procedure) Adverse Events(TEAEs). TEAEs are AEs with onset date on or after first dose of study intervention (placebo or MT10109L) in the pivotal study and ≤ 30 days after the study exit visit in the extension study.
Time Frame: Baseline to Day 720 or Study exit
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/MT10109L Dose 1 | Placebo/MT10109L Dose 2 | Placebo/MT10109L Dose 1 + Dose 2 | MT10109L Dose 1/Dose 1 | MT10109L Dose 2/Dose 2 | MT10109L Dose 1/Dose 1+2 | MT10109L Dose 2/Dose 1+2 | MT10109L Dose 1+2/Dose 1+2
Number analyzed (Participants) | 55 | 56 | 118 | 116 | 108 | 128 | 123 | 253
Participants | 18 | 4 | 31 | 34 | 11 | 22 | 42 | 73

3. Primary Outcome: Mean Change From Baseline in Pulse Rate (Beats Per Minute)
Description: The outcome reported here is the mean change in pulse rate from baseline to study exit.
Time Frame: Baseline to Day 720 or Study Exit
Population: All safety analyses were carried out using the ITT population, which was defined as all participants who enrolled in Study MT10109L-004 and received at least 1 intervention (MT10109L or placebo) in their prior Phase 3 study (MT10109L-001, -002, -005, or -006) or in the current study. The final outcome measure data reported here are the mean change measured among the participants at day 720 or study exit.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo/MT10109L Dose 1 | Placebo/MT10109L Dose 2 | Placebo/MT10109L Dose 1 + Dose 2 | MT10109L Dose 1/Dose 1 | MT10109L Dose 2/Dose 2 | MT10109L Dose 1/Dose 1+2 | MT10109L Dose 2/Dose 1+2 | MT10109L Dose 1+2/Dose 1+2
Number analyzed (Participants) | 55 | 56 | 118 | 116 | 108 | 128 | 123 | 253
beats/min | 3.2 (15.01) | -2.2 (13.35) | -1.2 (10.95) | 2.0 (12.77) | 0.6 (11.58) | 0.7 (10.97) | 3.0 (10.34) | 1.0 (8.93)

4. Primary Outcome: Mean Change From Baseline in Systolic Blood Pressure (mm Hg)
Description: The outcome reported here is the mean change in Systolic BP from baseline to study exit.
Time Frame: Baseline to Day 720 or Study Exit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo/MT10109L Dose 1 | Placebo/MT10109L Dose 2 | Placebo/MT10109L Dose 1 + Dose 2 | MT10109L Dose 1/Dose 1 | MT10109L Dose 2/Dose 2 | MT10109L Dose 1/Dose 1+2 | MT10109L Dose 2/Dose 1+2 | MT10109L Dose 1+2/Dose 1+2
Number analyzed (Participants) | 55 | 56 | 118 | 116 | 108 | 128 | 123 | 253
mmHg | 1.4 (12.59) | -1.9 (10.44) | 1.9 (14.44) | 0.6 (16.72) | 1.1 (13.84) | 1.8 (15.24) | 1.4 (14.17) | -0.4 (13.83)

5. Primary Outcome: Mean Change From Baseline in Diastolic Blood Pressure (mm Hg)
Description: The outcome reported here is the mean change in Diastolic BP from baseline to study exit.
Time Frame: Baseline to Day 720 or Study Exit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo/MT10109L Dose 1 | Placebo/MT10109L Dose 2 | Placebo/MT10109L Dose 1 + Dose 2 | MT10109L Dose 1/Dose 1 | MT10109L Dose 2/Dose 2 | MT10109L Dose 1/Dose 1+2 | MT10109L Dose 2/Dose 1+2 | MT10109L Dose 1+2/Dose 1+2
Number analyzed (Participants) | 55 | 56 | 118 | 116 | 108 | 128 | 123 | 253
mmHg | 1.1 (11.3) | -0.6 (11.75) | 1.3 (9.61) | 1.5 (11.68) | 0.7 (7.57) | 0.0 (10.62) | 2.3 (9.53) | -0.3 (9.46)

6. Primary Outcome: Mean Change From Baseline in Respiratory Rate (Breaths Per Minute)
Description: The outcome reported here is the mean change in respiratory rate from baseline to study exit.
Time Frame: Baseline to Day 720 or Study Exit
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo/MT10109L Dose 1 | Placebo/MT10109L Dose 2 | Placebo/MT10109L Dose 1 + Dose 2 | MT10109L Dose 1/Dose 1 | MT10109L Dose 2/Dose 2 | MT10109L Dose 1/Dose 1+2 | MT10109L Dose 2/Dose 1+2 | MT10109L Dose 1+2/Dose 1+2
Number analyzed (Participants) | 55 | 56 | 118 | 116 | 108 | 128 | 123 | 253
breaths/min | 0.3 (2.09) | 0.6 (2.15) | -0.5 (1.92) | 0.2 (2.78) | 0.5 (1.94) | -0.4 (2.29) | 0.4 (2.21) | -0.1 (2.3)

7. Primary Outcome: Number of Participants With Binding and Neutralizing Antibodies
Description: Only samples that tested positive in the binding antibody confirmatory assay were evaluated for neutralizing antibodies. The participants with positive neutralizing antibodies are only shown.
Time Frame: Baseline to Day 720 or Study Exit
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo/MT10109L Dose 1 | Placebo/MT10109L Dose 2 | Placebo/MT10109L Dose 1 + Dose 2 | MT10109L Dose 1/Dose 1 | MT10109L Dose 2/Dose 2 | MT10109L Dose 1/Dose 1+2 | MT10109L Dose 2/Dose 1+2 | MT10109L Dose 1+2/Dose 1+2
Number analyzed (Participants) | 55 | 56 | 118 | 116 | 108 | 128 | 123 | 253
Participants | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: The safety analyses were conducted in the Intent-to-Treat (ITT) population. All adverse events were collected from the signing of the ICF to 30 days after the participant's last study visit (Day 720/or early exit). Unless otherwise noted, safety results refer to TEAEs.
Description: An AE was considered a TEAE if:
  * The AE began on or after the date of the first dose of study intervention (lead-in or current study)
  * The AE was present before the date of the first dose of study intervention in this current study but increased in severity or became serious on or after the date of the first dose of study intervention in the current study.
Arm/Group | Placebo/MT10109L Dose 1 | Placebo/MT10109L Dose 2 | Placebo/MT10109L Dose 1 + Dose 2 | MT10109L Dose 1/Dose 1 | MT10109L Dose 2/Dose 2 | MT10109L Dose 1/Dose 1+2 | MT10109L Dose 2/Dose 1+2 | MT10109L Dose 1+2/Dose 1+2
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/56 | 0/118 | 2/116 | 0/108 | 0/128 | 0/123 | 0/253
Serious Adverse Events (participants affected / at risk) | 3/55 | 1/56 | 10/118 | 8/116 | 9/108 | 7/128 | 13/123 | 13/253
Other Adverse Events (participants affected / at risk) | 26/55 | 23/56 | 58/118 | 54/116 | 45/108 | 50/128 | 60/123 | 128/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/MT10109L Dose 1 (N=55) | Placebo/MT10109L Dose 2 (N=56) | Placebo/MT10109L Dose 1 + Dose 2 (N=118) | MT10109L Dose 1/Dose 1 (N=116) | MT10109L Dose 2/Dose 2 (N=108) | MT10109L Dose 1/Dose 1+2 (N=128) | MT10109L Dose 2/Dose 1+2 (N=123) | MT10109L Dose 1+2/Dose 1+2 (N=253)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basosquamous carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial spreading melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion induced (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo/MT10109L Dose 1 (N=55) | Placebo/MT10109L Dose 2 (N=56) | Placebo/MT10109L Dose 1 + Dose 2 (N=118) | MT10109L Dose 1/Dose 1 (N=116) | MT10109L Dose 2/Dose 2 (N=108) | MT10109L Dose 1/Dose 1+2 (N=128) | MT10109L Dose 2/Dose 1+2 (N=123) | MT10109L Dose 1+2/Dose 1+2 (N=253)
Injection site pain (General disorders) | 8 (8) | 0 (0) | 10 (10) | 17 (17) | 0 (0) | 8 (8) | 17 (17) | 23 (23)
Headache (Nervous system disorders) | 12 (12) | 1 (1) | 11 (11) | 12 (12) | 5 (5) | 13 (13) | 13 (13) | 27 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 6 (6) | 2 (2) | 2 (2) | 3 (3) | 4 (4) | 5 (5)
Hypertension (Vascular disorders) | 4 (4) | 2 (2) | 3 (3) | 5 (5) | 3 (3) | 3 (3) | 6 (6) | 9 (9)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 8 (8) | 3 (3) | 0 (0) | 4 (4) | 12 (12) | 20 (20)
Injection site haemorrhage (General disorders) | 1 (1) | 3 (3) | 8 (8) | 0 (0) | 6 (6) | 2 (2) | 7 (7) | 11 (11)
COVID-19 (Infections and infestations) | 7 (7) | 12 (12) | 22 (22) | 18 (18) | 31 (31) | 20 (20) | 22 (22) | 47 (47)
Nasopharyngitis (Infections and infestations) | 6 (6) | 4 (4) | 15 (15) | 9 (9) | 8 (8) | 9 (9) | 17 (17) | 31 (31)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 11 (11) | 6 (6) | 5 (5) | 7 (7) | 5 (5) | 15 (15)
Sinusitis (Infections and infestations) | 2 (2) | 5 (5) | 4 (4) | 3 (3) | 4 (4) | 3 (3) | 3 (3) | 7 (7)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Ligament Sprain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Procedural Pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
General research agreement between the sponsor and PI's that includes a confidentiality section that includes a statement that the sponsor is and shall remain the exclusive owner of 'Information'. 'Information' shall include, but shall not be limited to, protocols, trade secrets, know-how, formulations, inventions, techniques, equipment, data and results.

DOCUMENTS (2):
  • Study Protocol (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT04157686/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/86/NCT04157686/SAP_001.pdf